CLINICAL TRIAL: NCT05228288
Title: Conventional vs. Video-Assisted Laryngoscopy for Perioperative Endotracheal Intubation
Acronym: COVALENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University Hospital, Aachen (Other); University Hospital, Bonn (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COVALENT
Record Dates: First submitted 2022-02-07; First posted 2022-02-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Endotracheal Intubation
Keywords: anesthesiology; laryngoscopy; video-assisted laryngoscopy; intubation; airway management; patient safety; human factors; conventional laryngoscopy

STUDY DESIGN:
Intervention Model Description: In this randomized, controlled, three-armed parallel group design, multi-center trial, a total of more than 2500 adult patients scheduled for perioperative endotracheal intubation will be randomized. In equally large arms, video-assisted laryngoscopy with a Macintosh-shaped or a hyperangulated blade will be compared to the standard of care (direct laryngoscopy with Macintosh blade).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and data analysts will be blinded regarding the assignment of interventions.
  The randomization result will be communicated to the care providers non-verbally without revealing the result to the patient. Before data evaluation, the identifying variables will be made illegible. Investigators and care providers carrying out the intervention cannot be blinded due to the nature of the study. In the follow-up period two hours after the end of anesthesia, the outcome survey should be performed, if possible, by an investigator who was not involved in the intervention to ensure blinding. It will be documented whether blinding could be accomplished at this point. Un-blinding of the patient is only intended if an unexpected difficult airway situation occurred and the patient is issued a personal anaesthesia problem card. However, even in such cases, blinding can usually be ensured until after the last study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CDL (Active Comparator): Conventional direct laryngoscopy using a Macintosh blade
  Interventions: Procedure: Conventional direct laryngoscopy (CDL)
- M-VAL (Experimental): Video assisted laryngoscopy with a Macintosh-shaped blade
  Interventions: Procedure: Video assisted laryngoscopy with Macintosh-shaped blade (M-VAL)
- H-VAL (Experimental): Video assisted laryngoscopy with a hyper-angulated blade
  Interventions: Procedure: Video assisted laryngoscopy with hyper-angulated blade (H-VAL)

INTERVENTIONS:
Procedure: Conventional direct laryngoscopy (CDL) — This procedure is considered the gold standard for endotracheal intubation and is routinely used in the peri-operative setting as well as in intensive care and emergency medicine.
  Other Names: conventional direct laryngoscopy; conventional laryngoscopy
  Arms: CDL
Procedure: Video assisted laryngoscopy with Macintosh-shaped blade (M-VAL) — This device is implemented in most german hospitals and used when conventional direct laryngoscopy is not sufficient. By positioning the camera at the tip of the blade, the achievable field of view onto the glottic plane is improved.
  Other Names: video assisted laryngoscopy with Macintosh-shaped blade
  Arms: M-VAL
Procedure: Video assisted laryngoscopy with hyper-angulated blade (H-VAL) — The hyper-angulated blades are often used as a backup instrument when a view of the glottic plane cannot be achieved with the Macintosh blade due to anatomic abnormalities, even with a video-assisted laryngoscope.
  Other Names: video assisted laryngoscopy with hyper-angulated blade
  Arms: H-VAL

SUMMARY:
COVALENT is a randomized, controlled, multi-center study that aims to evaluate the clinical routine practice of endotracheal intubation in an operative setting comparing video-assisted laryngoscopy to direct laryngoscopy.

DETAILED DESCRIPTION:
Data on the routine use of video-assisted laryngoscopy in peri-operative intubations are rather inconsistent and ambiguous, in part due to small study populations and non-uniform outcome measures in past trials. Failed or prolonged intubation procedures are a reason for relevant morbidity and mortality. This study aims to determine whether video-assisted laryngoscopy (irrespective of the shape of the blade) is non-inferior to the standard method of direct laryngoscopy with respect to the first-pass success rate. Furthermore, validated tools from the field of human factors will be applied to examine within-team communication and task load during this critical medical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult, legally competent patients
* Scheduled for elective, non-cardiac surgical procedure
* Need for endotracheal intubation as determined during the premedication visit
* Informed consent
* Care providers performing the intubation have at least one year of training in anesthesiology and experience in the use of VAL

Exclusion Criteria:

* Lack of ability to give consent
* Previous participation in this study
* Pregnancy
* Need for fiberoptic intubation
* Patients scheduled for bariatric surgery
* Any circumstance that will lead the anesthesiologist(s) in charge to believe that random assignment of a laryngoscopy instrument may compromise patient safety during induction of anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2855 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Successful intubation | During the period of intubation (as soon as the laryngoscope blade passes the teeth row of the patient until the first capnographic end-expiratory carbon dioxide [CO2] detection is possible)
  The primary endpoint is the successful intubation at first attempt as a dichotomous (successful/unsuccessful) event. The first attempt begins with the laryngoscope spatula passing the patient's row of teeth. The attempt is considered unsuccessful if a complete retraction of the laryngoscope or the endotracheal tube from the oropharynx is necessary for any reason (need for bag ventilation, change of device, change of patient position, change in the curvature of the stylet, etc.). Maneuvers that can be performed during laryngoscopy, such as BURP (backward, upward, rightward pressure) or reclining the head, which end with successful intubation, count towards the first attempt.

SECONDARY OUTCOMES:
Parameters regarding the duration of the intervention | During the period of intubation (as soon as the laryngoscope blade passes the teeth row of the patient until the first capnographic end-expiratory CO2 detection is possible)
  Time to intubation and time to glottis view (as announced by the anesthesist)
Cormack & Lehane grade | During the period of intubation (as soon as the laryngoscope blade passes the teeth row of the patient until the first capnographic end-expiratory CO2 detection is possible)
  Grade 1 (full view of glottis), Grade 2a (partial view of glottis), Grade 2b (view only of posterior extremity of glottis or arytenoid cartilages), Grade 3 (view of epiglottis, none of the glottis), Grade 4 (neither view of glottis nor epiglottis)
Intubation success | During the period of intubation (as soon as the laryngoscope blade passes the teeth row of the patient for the first time until the first capnographic end-expiratory CO2 detection is possible)
  Total number of attempts. Number of attempts using the randomized device. Success rate of intubation attempts regarding the respective device.
Influence of the device on human factors during the intervention | During the period of intubation and maintenance of anesthesia
  Mayo High Performance Teamwork Scale, NASA-TLX (National Aeronautics and Space Administration's Task Load Index)
Complications: occurrence of one or more of the following | During the period of intubation (as soon as the laryngoscope blade passes the teeth row of the patient for the first time until the first capnographic end-expiratory CO2 detection is possible)
  Drop of SpO2 (oxygen saturation) below 90%. Regurgitation as announced by the anesthetist. Need for bronchoscopy due to suspected aspiration. Dental injury or dental clicks upon contact with the blade. Soft tissue injuries as detected by blood on the blade. Visible swelling. Bleeding or other injury of the lips. Need for resuscitation (administration of adrenalin, chest compressions, defibrillation or any combination thereof). Death. Occurence of any adverse event (AE) or serious adverse event (SAE).
Need for auxiliary devices or switch of laryngoscopy device | During the period of intubation (as soon as the laryngoscope blade passes the teeth row of the patient for the first time until the first capnographic end-expiratory CO2 detection is possible)
  Manœuvres to optimize intubation conditions after the first attempt at intubation has started. Switch to alternate laryngoscopy device. Switch of the anesthetists. Switch of airway device
Relevant vital parameters during the intervention | During the period of intubation (as soon as the laryngoscope blade passes the teeth row of the patient for the first time until the first capnographic end-expiratory CO2 detection is possible)
  Baseline SpO2 and lowest SpO2
Post-operative sore throat, coughing or hoarseness | End of surgery until two hours after the end of surgery
  Post-operative sore throat, coughing or hoarseness, according to the "Scoring System for Sore Throat, Cough, and Hoarseness" by Park et al. This outcome will not be assessed in patients who continue to be invasively ventilated > 2 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Schmid, MD, PhD, Principal Investigator — Department of Anaesthesiology, Medical Faculty Würzburg
Locations (1):
- University Hospital Wuerzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park SY, Kim SH, Lee AR, Cho SH, Chae WS, Jin HC, Lee JS, Kim YI. Prophylactic effect of dexamethasone in reducing postoperative sore throat. Korean J Anesthesiol. 2010 Jan;58(1):15-9. doi: 10.4097/kjae.2010.58.1.15. Epub 2010 Jan 31. PMID 20498806
- [Derived] Schmid B, Eckert D, Meixner A, Pistner P, Malzahn U, Berberich M, Happel O, Meybohm P, Kranke P. Conventional versus video-assisted laryngoscopy for perioperative endotracheal intubation (COVALENT) - a randomized, controlled multicenter trial. BMC Anesthesiol. 2023 Apr 18;23(1):128. doi: 10.1186/s12871-023-02083-3. PMID 37072702
- See also: covalent Website — https://covalent-trial.org/